CLINICAL TRIAL: NCT05876832
Title: Phase 3 Open-label, Multicenter, Randomized Study of XY0206 Versus Salvage Chemotherapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) With FMS-like Tyrosine Kinase 3(FLT3)-Internal Tandem Duplication（ITD） Mutation
Brief Title: A Study of XY0206 Versus Salvage Chemotherapy In Patients With Relapsed or Refractory AML With FLT3-ITD-Mutation (ALIVE)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XY0206AML3001
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XY0206 (Experimental): XY0206 will be administered orally once a day in continuous 28-day cycles.
  Interventions: Drug: XY0206
- Salvage chemotherapy (Active Comparator): Participants will receive salvage chemotherapy in 28-day cycles. Participants on Low-Dose Cytarabine (LoDAC) received 20 mg of cytarabine twice daily by subcutaneous (SC) injection for 10 days. Participants on azacitidine will receive 75 mg/m^2 daily by SC or IV injection for 7 days.Participants on fludarabine, cytarabine and granulocyte colony-stimulating factor (G-CSF) (FLAG) will receive 30 mg/m^2 of fludarabine daily by IV for 5 days (day 2 to 6), 1~2 g/m2 of cytarabine daily by IV for 5 days (day 2 to 6), and 300 μg/m^2 of G-CSF daily by SC or IV for 5 days (days 1 to 5). After completion of chemotherapy, G-CSF will be administered continually until absolute neutrophil count(ANC)>0.5 x 10^9 / L. Participants on mitoxantrone, etoposide, cytarabine(MEC) will receive 8 mg/m^2 of mitoxantrone daily by IV for 3 days (day 1 to 3), 100 mg/m2 of etoposide daily by IV for 7 days (day 1 to 7), and 100 mg/m^2 of cytarabine daily by IV for 7 days (days 1 to 7)
  Interventions: Drug: Salvage Chemotherapy

INTERVENTIONS:
Drug: XY0206 — Dosage form:Tablet;Multiple dose phase:Take the medicine once a day,37.5mg at a time.4 weeks of continuous medication is one course of treatment. After the first course of treatment, the subjects can continue to receive the experimental drug treatment until the subjects meet the withdrawal criteria.
  Arms: XY0206
Drug: Salvage Chemotherapy — Low-dose Cytarabine (LoDAC) or azacitidine, fludarabine, cytarabine and granulocyte colony-stimulating factor (FLAG) or mitoxantrone, etoposide, cytarabine (MEC)will be administered by subcutaneous (SC) and/or intravenous (IV) injections.
  Arms: Salvage chemotherapy

SUMMARY:
The purpose of this study is to determine the clinical benefit of XY0206 therapy in participants with FLT3-ITD mutated AML who are refractory to or have relapsed after prior AML therapy as shown with overall survival (OS) compared to salvage chemotherapy. In addition, this study is also to investigate the efficacy of XY0206 as assessed by CR/CRh rate in these subjects。

DETAILED DESCRIPTION:
Participants considered an adult according to local regulations at the time of signing informed consent will be randomized in a 2:1 ratio to receive XY0206 or salvage chemotherapy. Participants will enter the screening period up to 14 days prior to the start of treatment. Prior to randomization, the investigator will preselect a salvage chemotherapy regimen for each participant; options will include low-dose cytarabine (LoDAC),azacitidine, fludarabine, cytarabine and granulocyte colony-stimulating factor (FLAG) or mitoxantrone, etoposide and cytarabine (MEC) . The randomization will be stratified by remission from previous treatment and preselected salvage chemotherapy. Participants will be administered treatment over continuous 28-day cycles.

Participants who have a donor identified and with complete remission after treatment may undergo hematopoietic stem cell transplant (HSCT) without leaving the study.

After treatment discontinuation, participants will have a end-of-treatment visit within 7 days after treatment discontinuation, followed by a 30-day follow-up for safety. After that, long term follow-up will be done every 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old.
2. Subject has a diagnosis of primary AML or AML secondary to myelodysplastic syndrome (MDS) according to World Health Organization (WHO) classification as determined by pathology review at the treating institution.
3. Subject is refractory to or relapsed after prior AML therapy (with or without hematopoietic stem cell transplant ):

   * Advanced relapse after first-line AML therapy is defined as: the patients achieved Complete remission without minor residual diseases/complete remission/complete remission with partial hematologic recovery/complete remission with incomplete hematologic recovery/complete remission with incomplete platelet recovery/Morphologic leukemia- free state(CRMRD-/CR/CRh/CRi/CRp/MLFS )after first-line treatment and relapsed after 12 months with hematological relapse;
   * Patients with relapsed / refractory AML.
   * Refractory to first-line AML therapy is defined as:the patient did not achieve CRMRD-/CR/CRh/CRi/CRp/MLFS under initial therapy.A subject eligible for standard therapy must receive at least 1 cycle of an anthracycline containing induction block in standard dose for the selected induction regimen. A subject not eligible for standard therapy must have received at least 1 complete block of induction therapy seen as the optimum choice of therapy to induce remission for this subject.
   * Early relapse:Relapse within 12 months after consolidation therapy after achieving CRMRD-/CR/CRh/CRi/CRp/MLFS.
   * Relapse after 12 months but nonresponse to conventional chemotherapy after achieving CRMRD-/CR/CRh/CRi/CRp/MLFS.
   * Second or more relapse.
   * Patients who cannot tolerate intensive chemotherapy develop disease progression during continuous treatment with low-intensity drugs.
   * Persistence of extramedullary leukemia.
4. Patient is positive for FLT3-ITD mutation in bone marrow or whole blood.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Expected survival ≥12 weeks .
7. Patient must meet the following criteria as indicated on the clinical laboratory tests:

   * Serum creatinine ≤ 1.5 x ULN or an estimated glomerular filtration rate of ≥50 mL/min .
   * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
   * Serum total bilirubin (TBL) ≤ 1.5 x ULN.
   * Fridericia's Heart Rate Correction Formula (QTcF) interval ≤480 msec.
8. Female patients of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first study drug administration.Female patients of childbearing potential and male must be surgically sterile or willing to use highly effective birth control upon enrollment, during the treatment period, and for 6 months following the last dose of investigational drug.
9. The subject should be willing to provide evidence of valid diagnosis before treatment or undergo bone marrow puncture or biopsy for diagnosis, and receive bone marrow puncture or biopsy for efficacy evaluation after treatment.
10. Patients volunteered to participate in this study and signed the informed consent form.

Exclusion Criteria:

1. Patient was diagnosed as acute promyelocytic leukemia (APL), or Philadelphia chromosome（BCR-ABL）-positive leukemia (chronic myelogenous leukemia in blast crisis).
2. Patients who received live vaccine (including live attenuated vaccine) within 4 weeks before randomization and/or planed to receive live vaccine after enrollment.
3. Presence of FLT3-tyrosine kinase domain(TKD) mutation.
4. Patients were prior failed adequate treatment with FLT3 inhibitors.
5. AML with Central Nervous System Leukemia.
6. Patient has AML secondary to prior chemotherapy for other neoplasms, except for MDS.
7. Patients with other malignant tumors past or present,unless whose Disease-free survival period≥5 years.Non-melanin skin cancer, carcinoma in situ, or cervical intraepithelial neoplastic lesions with completed radical treatment (regardless of disease-free survival),and subjects with prostate cancer confined to the prostate and with no evidence of disease recurrence or progression,if they have started hormonal therapy or have undergone surgery to remove the malignancy or have undergone radical radiotherapy,will be eligible for the study.
8. Pretrial treatment conditions:

   * Patients who received hematopoietic stem cell transplantation within the 2 months before enrollment,or having clinically significant graft-versus-host disease (GVHD) or receiving systemic cortisol hormone therapy for GVHD.
   * Patients who received chemotherapy, biological therapy, targeted anti-tumor therapy within 14 days before the first use of the drug in this study or within 5 half-lives of the drug, or radiation therapy within 28 days.
   * Patients who participated in other clinical trials and received trial drugs within 28 days to the first study dose.
   * Patients who have had major surgery or significant traumatic injury within 28 days to the first study dose or planted to require major surgery during study treatment.
9. Concurrent disease conditions:

   * Patients are hepatitis B surface antigen or core antibody actives positive,and hepatitis B virus(HBV) DNA ≥2000IU/mL or 1×104 copy/mL.
   * Patients are hepatitis C virus (HCV) antibody actives positive and HCV-RNA quantification is above the upper limit of normal at each center.
   * Human immunodeficiency virus (HIV) seropositivity.
   * Patient has clinically obvious gastrointestinal abnormalities that may affect the intake, transport, or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc),patients with total gastrectomy or major gastrectomy (Billroth II), patients with a clear gastrointestinal bleeding tendency,or major gastrointestinal bleeding considered possible by the investigator.
   * Patient has uncontrolled epilepsy history.
   * Patient has uncontrolled hypertension defined as systolic blood pressure greater than 160 mmHg or diastolic pressure greater than 100 mmHg, despite optimal medical management and optimal measurement.
   * Patient has clinically significant abnormal serum lipase or amylase indicators during screening.
   * Patient has refractory intractable hypokalemia or hypomagnesemia.
   * Patient has clinically significant abnormality of coagulation profile, such as disseminated intravascular coagulation (DIC), hemophilia.
   * Patient has congestive heart failure New York Heart Association (NYHA) class 3 or 4 or patient with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram performed within 1 month before study entry results in a left ventricular ejection fraction that is ≥ 45%.
   * Patients with second degree (Mobitz II) or third degree atrioventricular block disease (except for patients who use the pacemaker) or complete left bundle branch block.
   * Patients with new clinically significant arrhythmias (except for sinus tachycardia caused by anemia, infection and AML) or patients with previous arrhythmias that require long-term use of drugs with QT-prolonging effects.
   * Patients with any one of the following diseases within 6 months prior to randomization:myocardial infarction,unstable angina pectoris,Patients undergoing coronary artery bypass graft(CABG) or peripheral artery bypass implantation,congestive heart-failure,Cerebrovascular events (including cerebral hemorrhage and cerebral infarction, etc.),Deep venous thrombosis (except for deep venous thrombosis due to peripherally inserted central venous catheter (PICC) catheterization),pulmonary embolism and other diseases that the researcher considers inappropriate to participate in this study.
   * Patients with diagnosed or suspected long QT syndrome at screening (including a family history of long QT syndrome).
   * Patient has an active uncontrolled infection.
   * Patient has severe unhealed wounds, ulcers, or fractures.
   * Females who are pregnant or breastfeeding.
   * Patients are not suitable for the study in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Interim analysis: Complete remission(CR)/CR with partial hematologic recovery(CRh) rate in the experimental group. | up to 3 years.
  The complete remission and complete remission with partial hematological recovery (CR/CRh) rate was defined as the number of subjects who achieved either CR or CRh at any of the postbaseline visits divided by the number of subjects in the analysis population.
The final analysis: Overall Survival(OS). | up to 3 years .
  Overall survival was defined as the time from the date of randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Key secondary end point: Event-Free Survival (EFS). | up to 3 years.
  Event-free survival (EFS) is defined as the time from the date of randomization until the date of documented relapse， treatment failure or death whichever occurs first.
Key secondary end point: CR/CRh rate . | up to 3 years.
  The CR/CRh rate was defined as the number of subjects who achieved either CR or CRh at any of the postbaseline visits divided by the number of subjects in the analysis population.
CR rate. | up to 3 years.
  The CR rate was defined as the number of subjects who achieved the best response of CR divided by the number of subjects in the analysis population.
Duration of remission (DOR). | up to 3 years.
  Duration of remission included duration of composite complete remission (CRc), duration of complete remission (CR)/ complete remission with partial hematologic recovery (CRh), duration of CRh, duration of CR and duration of response (CRc + partial remission (PR).
Composite complete remission rate. | up to 3 years.
  CRc rate is defined as the remission rate of all CR, CRh , CR with incomplete hematologic recovery(CRi) or Morphologic leukemia- free state(MLFS).
minimal residual disease(MRD) negative rate | up to 3 years.
  MRD negative rate is defined as the percentage of participants without MRD.
Time to remission(TTR). | up to 3 years.
  Time to remission(TTR) is defined as the time from the date of randomization until the date of is defined as the time from the date of randomization until the date of remission.
Transplantation rate. | up to 3 years.
  Transplantation rate is defined as the percentage of participants undergoing hematopoietic stem cell transplant (HSCT).
Safety assessed by adverse events. | up to 3 years.
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment.
Population pharmacokinetic of XY0206. | Cycle 1 Day 15: predose and up to 4 hours post-dose; Day 28 predose of subsequent cycles. A cycle is 28 days.
  Observed trough concentration (Ctrough).

IPD SHARING:
Plan to Share IPD: No